CLINICAL TRIAL: NCT04699292
Title: International Prospective Registry on Local Treatment Approaches in Myxoid Liposarcomas
Brief Title: International Prospective Registry on Local Treatment Approaches in MLS
Status: Recruiting | Type: Observational
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Radboud University Medical Center (Other); Maastro Clinic, The Netherlands (Other); University Medical Center Groningen (Other); Leiden University Medical Center (Other); Vienna General Hospital (Other); M.D. Anderson Cancer Center (Other); University Hospital, Antwerp (Other); Universitetssykehus (Unknown); Haukeland University Hospital (Other); Universitäts-Frauenklinik Graz (Other); University Hospital Heidelberg (Other); Mayo Clinic (Other); Aarhus University Hospital (Other); National Cancer Center, Japan (Other Government); Princess Margaret Hospital, Canada (Other); MOUNT SINAI HOSPITAL (Other); University of Sydney (Other); Institute for Cancer Research and treatment (Unknown); Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other); Institut Curie (Other); Australia and New Zealand Sarcoma Association (Other)
Responsible Party: Sponsor
Other Study IDs: M20DMY; IRBd20-354 (Other: The Netherlands Cancer Institute)
Record Dates: First submitted 2021-01-06; First posted 2021-01-07 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Myxoid Liposarcoma
MeSH Terms: conditions — Liposarcoma, Myxoid | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Cohort A: MLS patients managed by surgery only
  Interventions: Procedure: Surgery
- Cohort B: MLS patients receiving preoperative RT to a dose of 36 Gy (equivalent) followed by surgery
  Interventions: Procedure: Surgery; Radiation: Preoperative RT 36Gy
- Cohort C: MLS patients receiving preoperative RT to a dose of 50 Gy (equivalent) followed by surgery
  Interventions: Procedure: Surgery; Radiation: Preoperative RT 50Gy
- Cohort D: MLS patients receiving surgery followed by postoperative RT to a dose of 50-66 Gy (equivalent)
  Interventions: Procedure: Surgery; Radiation: Postoperative RT 50-66Gy
- Cohort E: MLS patients with oligometastatic and/or oligoprogressive disease receiving definitive RT to a dose of 36Gy (equivalent)
  Interventions: Radiation: RT 36Gy

INTERVENTIONS:
Procedure: Surgery — Surgery
  Groups: Cohort A; Cohort B; Cohort C; Cohort D
Radiation: Preoperative RT 36Gy — Preoperative radiotherapy to 36Gy (equivalent)
  Groups: Cohort B
Radiation: Preoperative RT 50Gy — Preoperative radiotherapy to 50Gy (equivalent)
  Groups: Cohort C
Radiation: Postoperative RT 50-66Gy — Postoperative radiotherapy to 50-66Gy (equivalent)
  Groups: Cohort D
Radiation: RT 36Gy — Definitive radiotherapy to 36Gy (equivalent)
  Groups: Cohort E

SUMMARY:
To prospectively study commonly used local treatment approaches in Myxoid Liposarcoma (MLS)

DETAILED DESCRIPTION:
In order to confirm the promising results of the 36 Gy dose level in the DOREMY trial (NCT02106312) and to compare outcome with other local treatment approaches.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Biopsy proven MLS, including the reciprocal chromosomal translocation t(12;16)(q13;p11)
* ECOG PS 0-2
* Written informed consent to share coded information in this international Registry

Exclusion Criteria:

* Prior radiotherapy to the target area
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Myxoid Liposarcoma (MLS) that will be treated in one of the participating Sarcoma Reference Centers according to one of the treatment approaches defined in the 5 cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-18 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival | From surgery to the end of at least 5 years of follow-up
  Survival from surgery to local recurrence (event) or last follow-up

SECONDARY OUTCOMES:
Wound complications | From surgery to 6 months of follow-up
  Any wound complication requiring intervention
Late toxicity | From 3 months after surgery to the end of at least 5 years of follow-up
  Any grade ≥2 late (radiation-induced) toxicity according to CTCAE v5.0 toxicity criteria

OTHER OUTCOMES:
Patient-Reported Outcome Measures (PROMs) | From baseline visit to the end of 5 years of follow-up
  PRO-CTCAE Item Library; relevant questions from the Patient-Reported Outcomes version of the CTCAE (PRO-CTCAE)
Health-Related Quality of Life (HRQoL) | From baseline visit to the end of 5 years of follow-up
  EORTC QLQ-C30; 30-item HRQoL questionnaire; EORTC Items Library; 3 questions to assess some radiotherapy-specific HRQoL; EQ5D-5L; descriptive system for measurement of health; iMCQ; relevant items from the Medical Consumption Questionnaire (iMCQ) to assess medical consumption; PRODISQ; PROductivity and DISease Questionnaire to assess all relevant aspects of the relationship between health and productivity;

CONTACTS AND LOCATIONS:
Overall Officials: Rick Haas, MD/PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- The Netherlands Cancer Institute, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: No